CLINICAL TRIAL: NCT02738333
Title: A Phase 3b, Multicenter, Randomized, Open-Label Study to Investigate the Efficacy and Safety of Ledipasvir/Sofosbuvir Fixed-Dose Combination for 12 Weeks in Subjects With Chronic Genotype 2 HCV Infection
Brief Title: Ledipasvir/Sofosbuvir Fixed-Dose Combination for 12 Weeks in Participants With Chronic Genotype 2 HCV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-1903
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Results first posted 2018-03-14 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-02

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination; Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- LDV/SOF (Cohort 1) (Experimental): LDV/SOF FDC for 12 weeks
  Interventions: Drug: LDV/SOF
- SOF+RBV (Cohort 1) (Experimental): SOF+RBV for 12 weeks
  Interventions: Drug: SOF; Drug: RBV
- LDV/SOF (Cohort 2) (Experimental): Participants who are ineligible for or intolerant to RBV therapy will receive LDV/SOF FDC for 12 weeks.
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: LDV/SOF — 90/400 mg FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977
  Arms: LDV/SOF (Cohort 1); LDV/SOF (Cohort 2)
Drug: SOF — 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
  Arms: SOF+RBV (Cohort 1)
Drug: RBV — Capsules administered orally in a divided daily dose according to package insert weight-based dosing recommendations (≤ 60 kg = 600 mg, > 60 kg to ≤ 80 kg = 800 mg, and > 80 kg = 1000 mg)
  Other Names: REBETOL®
  Arms: SOF+RBV (Cohort 1)

SUMMARY:
The primary objectives of this study are to evaluate the antiviral efficacy of therapy with ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) and to evaluate the safety and tolerability of LDV/SOF FDC and sofosbuvir (SOF) + ribavirin (RBV) in participants with chronic genotype 2 hepatitis C virus (HCV) infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic genotype 2 HCV-infected males and non-pregnant/non-lactating females
* Aged 20 years or older
* Treatment naive or treatment experienced
* At least 20 subjects will have Child-Pugh-A compensated cirrhosis. In Cohort 2, participants must be ineligible or intolerant of RBV.

Key Exclusion Criteria:

* Previous exposure to an NS5A or NS5B inhibitor
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Pregnant or nursing female or male with pregnant female partner

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (37):
- Japan (37):
  - Bunkyō City
  - Chiba
  - Chūō
  - Ehime
  - Fukuoka
  - Fukuyama
  - Gifu
  - Ibaraki
  - Ikeda
  - Iruma-gun
  - Izunokuni
  - Kagoshima
  - Kashihara
  - Kitakyushu
  - Kumamoto
  - Kyoto
  - Maebashi
  - Matsumoto
  - Morioka
  - Musashino
  - Nagasaki
  - Nagoya
  - Nishinomiya
  - Okayama
  - Osaka
  - Ōgaki
  - Ōmura
  - Saga
  - Sagamihara
  - Sapporo
  - Sendai
  - Suita
  - tabashi City
  - Takamatsu
  - Ube
  - Yamagata
  - Yufu

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Japan. The first participant was screened on 12 April 2016. The last study visit occurred on 11 May 2017.
Pre-assignment Details: 266 participants were screened.
Groups:
- LDV/SOF (Cohort 1): Ledipasvir/sofosbuvir (LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet once daily for 12 weeks
- SOF+RBV (Cohort 1): Sofosbuvir (SOF) 400 mg tablet once daily + ribavirin (RBV) capsules (600, 800, or 1000 mg daily based on weight) for 12 weeks
- LDV/SOF (Cohort 2): LDV/SOF (90/400 mg) FDC tablet once daily for 12 weeks in participants who are ineligible for or intolerant to RBV therapy
Period: Overall Study
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Started | 106 | 108 | 25
Completed | 104 | 108 | 25
Not Completed | 2 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who took at least 1 dose of study drug
Groups:
- LDV/SOF (Cohort 1): LDV/SOF (90/400 mg) FDC tablet once daily for 12 weeks
- SOF+RBV (Cohort 1): SOF 400 mg tablet once daily + RBV capsules (600, 800, or 1000 mg daily based on weight) for 12 weeks
- Total: Total of all reporting groups
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2) | Total
Number analyzed (Participants) | 106 | 108 | 25 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10.5) | 60 (12.3) | 74 (7.1) | 61 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 71 | 19 | 144
  Male | 52 | 37 | 6 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 106 | 108 | 25 | 239
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 106 | 108 | 25 | 239
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 88 | 86 | 15 | 189
    CT | 17 | 19 | 10 | 46
    TT | 1 | 3 | 0 | 4
HCV RNA (log10 IU/mL) [Mean (Standard Deviation); unit: log10 IU/mL] | 6.1 (0.79) | 6.1 (0.79) | 5.9 (0.72) | 6.0 (0.78)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 30 | 36 | 10 | 76
  ≥ 800,000 IU/mL | 76 | 72 | 15 | 163

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who were randomized and took at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 106 | 108 | 25
percentage of participants | 96.2 [90.6 to 99.0] | 95.4 [89.5 to 98.5] | 96.0 [79.6 to 99.9]
Statistical Analysis 1: Comparison: LDV/SOF (Cohort 1) vs SOF+RBV (Cohort 1); Test type: Non-Inferiority — A sample size of 100 participants per treatment group would provide over 90% power to establish non-inferiority in the SVR12 rates between the LDV/SOF group and SOF+RBV group. Sample size was based on the assumptions that the clinically meaningful non-inferiority margin is 10%, both groups have a SVR12 rate of 96%, and the significance level is 0.025 one-sided; Difference in proportions = 0.9, 95% CI 2-sided [-5.3 to 7.1] — Difference in proportions between treatment groups and associated 95% confidence intervals (CI) are calculated based on stratum-adjusted Mantel-Haenszel proportions

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 106 | 108 | 25
percentage of participants | 0.9 | 1.9 | 0

3. Secondary Outcome: Percentage of Participants With SVR at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 106 | 108 | 25
percentage of participants | 97.2 [92.0 to 99.4] | 98.1 [93.5 to 99.8] | 96.0 [79.6 to 99.9]

4. Secondary Outcome: Percentage of Participants With SVR at 24 Weeks After Discontinuation of Therapy (SVR24)
Description: SVR 24 was defined as HCV RNA < LLOQ at 24 weeks after stopping study treatment.
Time Frame: Posttreatment Week 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 106 | 108 | 25
percentage of participants | 96.2 [90.6 to 99.0] | 95.4 [89.5 to 98.5] | 96.0 [79.6 to 99.9]

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 1
Time Frame: Week 1
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 106 | 108 | 25
percentage of participants | 24.5 [16.7 to 33.8] | 31.5 [22.9 to 41.1] | 32.0 [14.9 to 53.5]

6. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 2
Time Frame: Week 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 106 | 107 | 25
percentage of participants | 73.6 [64.1 to 81.7] | 76.6 [67.5 to 84.3] | 76.0 [54.9 to 90.6]

7. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 3
Time Frame: Week 3
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 106 | 107 | 25
percentage of participants | 90.6 [83.3 to 95.4] | 90.7 [83.5 to 95.4] | 96.0 [79.6 to 99.9]

8. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 4
Time Frame: Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 106 | 107 | 25
percentage of participants | 98.1 [93.4 to 99.8] | 96.3 [90.7 to 99.0] | 100.0 [86.3 to 100.0]

9. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 5
Time Frame: Week 5
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 105 | 107 | 25
percentage of participants | 98.1 [93.3 to 99.8] | 99.1 [94.9 to 100.0] | 100.0 [86.3 to 100.0]

10. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 6
Time Frame: Week 6
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 105 | 107 | 25
percentage of participants | 99.0 [94.8 to 100.0] | 99.1 [94.9 to 100.0] | 100.0 [86.3 to 100.0]

11. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 8
Time Frame: Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 105 | 107 | 25
percentage of participants | 100.0 [96.5 to 100.0] | 100.0 [96.6 to 100.0] | 100.0 [86.3 to 100.0]

12. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 10
Time Frame: Week 10
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 105 | 107 | 25
percentage of participants | 100.0 [96.5 to 100.0] | 100.0 [96.6 to 100.0] | 100.0 [86.3 to 100.0]

13. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 12
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 105 | 106 | 25
percentage of participants | 100.0 [96.5 to 100.0] | 100.0 [96.6 to 100.0] | 100.0 [86.3 to 100.0]

14. Secondary Outcome: Change From Baseline in HCV RNA at Week 1
Time Frame: Baseline; Week 1
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 106 | 107 | 25
log10 IU/mL | -4.18 (0.540) | -4.34 (0.602) | -4.24 (0.550)

15. Secondary Outcome: Change From Baseline in HCV RNA at Week 2
Time Frame: Baseline; Week 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 106 | 107 | 25
log10 IU/mL | -4.76 (0.759) | -4.81 (0.772) | -4.64 (0.719)

16. Secondary Outcome: Change From Baseline in HCV RNA at Week 3
Time Frame: Baseline; Week 3
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 106 | 107 | 25
log10 IU/mL | -4.87 (0.780) | -4.89 (0.790) | -4.75 (0.714)

17. Secondary Outcome: Change From Baseline in HCV RNA at Week 4
Time Frame: Baseline; Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 106 | 107 | 25
log10 IU/mL | -4.89 (0.782) | -4.91 (0.794) | -4.76 (0.719)

18. Secondary Outcome: Change From Baseline in HCV RNA at Week 5
Time Frame: Baseline; Week 5
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 105 | 107 | 25
log10 IU/mL | -4.91 (0.781) | -4.92 (0.794) | -4.76 (0.719)

19. Secondary Outcome: Change From Baseline in HCV RNA at Week 6
Time Frame: Baseline; Week 6
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 105 | 107 | 25
log10 IU/mL | -4.91 (0.781) | -4.92 (0.793) | -4.76 (0.719)

20. Secondary Outcome: Change From Baseline in HCV RNA at Week 8
Time Frame: Baseline; Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 105 | 107 | 25
log10 IU/mL | -4.92 (0.785) | -4.93 (0.794) | -4.76 (0.719)

21. Secondary Outcome: Change From Baseline in HCV RNA at Week 10
Time Frame: Baseline; Week 10
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 105 | 107 | 25
log10 IU/mL | -4.92 (0.785) | -4.93 (0.794) | -4.76 (0.719)

22. Secondary Outcome: Change From Baseline in HCV RNA at Week 12
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 105 | 106 | 25
log10 IU/mL | -4.92 (0.785) | -4.92 (0.794) | -4.76 (0.719)

23. Secondary Outcome: Percentage of Participants With Overall Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
Number analyzed (Participants) | 106 | 108 | 25
percentage of participants | 2.8 | 3.7 | 4.0

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set: participants who took at least 1 dose of study drug
Arm/Group | LDV/SOF (Cohort 1) | SOF+RBV (Cohort 1) | LDV/SOF (Cohort 2)
All-Cause Mortality (participants affected / at risk) | 1/106 | 0/108 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/106 | 1/108 | 1/25
Other Adverse Events (participants affected / at risk) | 25/106 | 48/108 | 7/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF (Cohort 1) (N=106) | SOF+RBV (Cohort 1) (N=108) | LDV/SOF (Cohort 2) (N=25)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF (Cohort 1) (N=106) | SOF+RBV (Cohort 1) (N=108) | LDV/SOF (Cohort 2) (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 | 25 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 2 | 2
Pyrexia (General disorders) | 0 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 12 | 23 | 1
Headache (Nervous system disorders) | 10 | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (4):
  • Study Protocol: Original (2015-12-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT02738333/Prot_004.pdf
  • Study Protocol: Amendment 1 (2016-01-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT02738333/Prot_005.pdf
  • Study Protocol: Amendment 2 (2016-02-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT02738333/Prot_006.pdf
  • Statistical Analysis Plan (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT02738333/SAP_007.pdf